CLINICAL TRIAL: NCT02266693
Title: Efficacy of Transdiagnostic Internet-based CBT for Early Illness Unipolar Depression and Anxiety
Brief Title: Transdiagnostic iCBT for Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Arun Ravindran, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 057/2012
Record Dates: First submitted 2014-10-07; First posted 2014-10-17 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Major Depressive Disorder; Social Anxiety Disorder; Panic Disorder; Generalized Anxiety Disorder
Keywords: Cognitive Behavioural Therapy; Internet Based; CBT; Transdiagnostic; MDD; PD; SAD; GAD; iCBT
MeSH Terms: conditions — Depressive Disorder, Major; Phobia, Social; Panic Disorder; Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICBT Group (Experimental): The iCBT program consists of weekly online lessons, weekly homework assignments, regular automatic email reminders about lessons and homework, weekly contact via phone or email with a CBT therapist, and access to a large online library of written resources about depression and anxiety and application of CBT skills. The CBT therapist contacts all participants once a week to review lessons, assist patients with treatment difficulties, reinforce progress and encourage continued engagement with the program. Therapist-patient contact is limited to 10 minutes per patient per week.
  Interventions: Behavioral: iCBT
- Waitlist Group (No Intervention): Upon completion of the 8-week study wait-list period (i.e. their study participation), the opportunity to participate in iCBT, outside the study framework will be provided.

INTERVENTIONS:
Behavioral: iCBT — The iCBT program consists of weekly online lessons, weekly homework assignments, regular automatic email reminders about lessons and homework, weekly contact via phone or email with a CBT therapist, and access to a large online library of written resources about depression and anxiety and application of CBT skills. The CBT therapist contacts all participants once a week to review lessons, assist patients with treatment difficulties, reinforce progress and encourage continued engagement with the program. Therapist-patient contact is limited to 10 minutes per patient per week.
  Other Names: Internet based Cognitive Behavioural Therapy
  Arms: ICBT Group

SUMMARY:
This 8-week, pilot randomized, controlled trial to evaluate the benefits of transdiagnostic Internet-based CBT (iCBT) in young adults with MDD, SAD, PD or GAD. The investigators hypothesize that patients who receive iCBT will show significant improvement in anxiety symptoms and functioning, compared to a wait-list group. This pilot randomized controlled study will assess the efficacy of transdiagnostic iCBT in 60 young adults.

DETAILED DESCRIPTION:
Unipolar depression and anxiety disorders (particularly social anxiety disorder [SAD], generalized anxiety disorder [GAD] and panic disorder [PD]) are among the most common forms of mental illnesses. They often have a chronic course, and are frequently associated with co-morbidities, significant disability, and poor quality of life. Published epidemiologic studies indicate that these conditions typically emerge during early adolescence and adulthood, and are often poorly recognized, resulting in delay of several years before help is sought. Such delay is often attributed to the non-recognition of the significance of the symptoms, lack of information on or access to services, and embarrassment and fear of stigma, but each effective early treatment can reduce co-morbidities and improve prognosis.

Cognitive behaviour therapy (CBT) is recognized as the single most effective psychological intervention for depression and anxiety, but accessibility is affected by therapist costs and long wait times for OHIP-covered services. Internet-based CBT (iCBT) is an innovative alternative with higher accessibility and cost-efficiency than group CBT, but with comparable efficacy. Transdiagnostic models of iCBT that treat depression, SAD, PD and GAD within one program have shown efficacy in preliminary trials and may offer even greater accessibility and economy, as several depressed and anxious populations can be treated with the same protocol. As a non-pharmacological treatment option enhanced by technological advances, iCBT is likely to appeal to tech-savvy young adults. However, it has not been evaluated specifically in a young adult population, thus far.

This 8-week, multi-site, randomized, controlled trial to evaluate the benefits of trandiagnostic iCBT in 60 young adults with unipolar depression and/or SAD, PD or GAD. We hypothesize that patients who receive iCBT will show significant improvement in depressive and anxiety symptoms and functioning, compared to a wait-list group.

ELIGIBILITY:
Inclusion Criteria:

1. Age range (18-29 years).
2. Primary diagnosis of MDD, SAD, PD and/or GAD, per the DSM-IV-TR.
3. A score ≥17 on the first 17 items of the Hamilton Depression Rating Scale (HAM-D)55
4. A score ≥17 on the Hamilton Anxiety Rating Scale (HAM-A)56.
5. Score ≥50 on the Leibowitiz Social Anxiety Scale (LSAS),57 ≥10 on the Panic Disorder Severity Scale (PDSS)58 and/or ≥60 the Penn State Worry Questionnaire (PSWQ).59
6. Currently unmedicated or on stable and adequate doses of medication for at least 4 weeks.
7. Co-morbidities are allowed and will be documented.

Exclusion Criteria:

1. Primary diagnosis of any psychotic disorder or any other anxiety disorder (OCD, PTSD).

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2014-08; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HAM-D) Total Score | Baseline to study endpoint (Week 8)
Change in Hamilton Anxiety Rating Scale (HAM-A) Total Score | Baseline to study endpoint (Week 8)
Change in Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR) Total Score | Baseline to study endpoint (Week 8)
Change in Liebowitz Social Anxiety Scale (LSAS) Total Score | Baseline to study endpoint (Week 8)
Change in Panic Disorder Severity Scale Total Score | Baseline to study endpoint (Week 8)
Change in Penn State Worry Questionnaire Total Score | Baseline to study endpoint (Week 8)

SECONDARY OUTCOMES:
Change in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) Total Score | Baseline to study endpoint (Week 8)
Change in Sheehan Disability Scale (SDS) Total Score | Baseline to study endpoint (Week 8)
Change in Clinical Global Impression (CGI) | Baseline to study endpoint (Week 8)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Ravindran, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research